CLINICAL TRIAL: NCT02182440
Title: A DB Four-Arm, Parallel Group, Proof of Concept, Dose-Finding Adaptive Phase 2a/2b RCT to Investigate the Safety, Tolerability and Efficacy and Effect on QoL of Human Recombinant Alkaline Phosphatase in Patients With Sepsis-Associated AKI
Brief Title: A Safety, Tolerability, Efficacy and QoL Study of Human recAP in the Treatment of Patients With SA-AKI
Acronym: STOP-AKI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AM-Pharma (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-recAP-AKI-02-01; 2014-000761-40 (EudraCT Number)
Record Dates: First submitted 2014-06-27; First posted 2014-07-08 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Acute Kidney Injury
Keywords: SA-AKI; Sepsis; AKI; Recombinant Alkaline Phosphatase; recAP
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): 1 hour IV infusion once daily for 3 days
  Interventions: Other: Placebo
- 0.4 mg/kg (250 U/kg) recAP (Experimental): 1 hour IV infusion once daily for 3 days
  Interventions: Biological: recAP
- 0.8 mg/kg (500 U/kg) recAP (Experimental): 1 hour IV infusion once daily for 3 days
  Interventions: Biological: recAP
- 1.6 mg/kg (1000 U/kg) recAP (Experimental): 1 hour IV infusion once daily for 3 days
  Interventions: Biological: recAP

INTERVENTIONS:
Biological: recAP — One hour infusions once daily for three days
  Other Names: Recombinant Alkaline Phosphatase
  Arms: 0.4 mg/kg (250 U/kg) recAP; 0.8 mg/kg (500 U/kg) recAP; 1.6 mg/kg (1000 U/kg) recAP
Other: Placebo — 1 hour IV infusion once daily for 3 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether recombinant Alkaline Phosphatase (recAP) is effective and save, and to determine the most effective dose, in the treatment of patients with acute kidney injury caused by sepsis.

DETAILED DESCRIPTION:
Design:

Adaptive trial with two stages and interim analysis

* Stage 1: four arms; three dose groups and placebo. n=30/arm. (n=120)
* Interim analysis based on 120 subjects, with continued recruitment, adding 11 subjects to Stage 1 safety population (n=131): to evaluate safety and select dose for stage 2
* Stage 2: one dose group and placebo. N=85/arm. (n=170) Total n in the study: 301.

Primary objectives

* To investigate the effect of recAP on renal function (measured creatinine clearance D1-D7 period, incidence and duration of renal replacement therapy (RRT) over 28 days, eGFR at D60 and D90) and related clinical parameters (ICU stay, Hospital stay, Mechanical ventilation over 28 days, SOFA and SAPS2 scores 28 days) in patients with SA-AKI.
* To determine effective therapeutic dose(s) of recAP.

Secondary objectives

* To investigate the safety and tolerability of recAP in patients with SA AKI. (assessed by independent Data Monitoring Board, adverse events over 90 days study period, laboratory values, ECG, physical examniations, vital signs, Anti Drug Antibodies)
* To investigate the pharmacokinetic profile (PK) of recAP in a subset of patients (part 1, n=120) with SA AKI. (Population PK; AUC D1-7, Cmax, Cmin, Tmax, terminal T1/2)
* To investigate the immunogenic potential of recAP in patients with SA AKI. (anti-drug antibodies at D14, D28, D60 and D90)
* To investigate the effect on quality of life (using the EuroQol, EQ-5D) following study inclusion, at ICU discharge, and Day 90.

Other objectives

• To evaluate whether specific patient groups can be identified that benefit most from recAP treatment or patient groups that are non-responders

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (patient, legal representative or independent investigator)
2. Age 18 to 85 years, inclusive
3. Is admitted to the ICU or Intermediate Care Unit
4. Has diagnosis of sepsis (< 96 hrs prior to first study drug), according to criteria defined by the American College of Chest Physicians/Society of Critical Care Medicine:

   1. Has a proven or strongly suspected bacterial infection.
   2. Has at least 2 of 4 SIRS criteria 72 hrs < screening and 96 hrs < first study drug
5. First diagnosis of AKI: AKI Stage 1 or greater, according to the AKIN criteria (time-window adjusted):

   1. Increase in serum creatinine > 26.2 µmol/L (0.30 mg/dL) in 48 hrs prior to screening, or
   2. Increase in serum creatinine to > 150% (> 1.5-fold) from reference creatinine value in 48 hrs prior to screening
   3. Urinary output < 0.5 mL/kg/h for > 6 hours following adequate fluid resuscitation
6. Continuing AKI needs to be confirmed by a confirmative fluid corrected serum creatinine measure, or
7. When the AKI diagnosis was made according to the AKIN urine output criteria (urinary output < 0.5 mL/kg/h for > 6 hours), the oliguria or anuria should still meet the AKIN urine output criteria prior to randomization.

Exclusion Criteria:

1. Woman of childbearing potential with a positive pregnancy test, pregnant, or breastfeeding.
2. Weighs more than 115 kg (253 lb).
3. Has life support limitations.
4. Is known to be human immunodeficiency virus positive.
5. Has urosepsis.
6. Is already on dialysis (RRT) or anticipated to receive RRT within 24 hours after study drug dosing due to the underlying disease.
7. Is receiving immunosuppressant treatment or is on chronic high doses of steroids equivalent to prednisone/prednisolone 0.5 mg/kg/day, including solid organ transplant patients. Patients with septic shock treated with hydrocortisone (e.g., 3 × 100 mg) can be included.
8. Is expected to have rapidly fatal outcome (within 24 hours).
9. Has known, confirmed fungal sepsis.
10. Has advanced chronic liver disease, confirmed by a Child-Pugh score of 10 to 15.
11. Has acute pancreatitis with no established source of infection.
12. Has participated in another investigational study within 30 days prior to enrollment.
13. Is not expected to survive for 28 days due to medical conditions other than SA AKI, including cancer, end-stage cardiac disease, cardiac arrest requiring cardiopulmonary resuscitation or with pulseless electrical activity or asystole within the past 30 days, end stage lung disease, and end stage liver disease.
14. Has known prior history of Chronic Kidney Disease with a documented estimated Glomerular Filtration Rate (eGFR) < 60 mL/min by Modification of Diet in Renal Disease MDRD or CKD-EPI formula, known GFR < 60 mL/min, or a known history of persistent creatinine level > 150 µmol/L (1.70 mg/dL) for reasons other than the current sepsis condition.
15. Has diagnosis of malaria or other parasite infections.
16. Has burns on > 20% of body surface.
17. Has had AKI diagnosis according to inclusion criteria > 24 hours prior to study drug administration.
18. Is anticipated to be treated with non-continuous RRT from Day 1 to Day 7.
19. During Day 1 to Day 7 continuous RRT is anticipated to be started or stopped not according to per protocol criteria.
20. The AKI is most likely attributable to other causes than sepsis, such as nephrotoxic drugs and renal perfusion-related.
21. Improvement in serum creatinine of at least 0.30 mg/dL or (26.2 µmol/L) prior to administration of the study drug.
22. Patients who use nephrotoxic medication and who fulfill the SA-AKI inclusion criteria at screening are not eligible if the use of this nephrotoxic medication is to continue when alternative, medically appropriate, non-nephrotoxic medication is available.
23. Has a history of known IV drug abuse.
24. Is an employee or family member of the investigator or study site personnel.
25. Has active hematological malignancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Arend, MD DiMD, Study Director — AM Pharma BV; Peter Pickkers, Prof MD. PhD, Study Chair — Department Intensive Care, Radboud University Medical Center
Locations (58):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Tampa General Hospital, Division Emergency Medicine, Tampa, Florida
  - Eastern Idaho Medical Consultants LLC, Idaho Falls, Idaho
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - UPMC, Pittsburgh, Pennsylvania
  - University of Texas Houston Medical School, Houston, Texas
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Universitätsklinik für Allgemeine und Chirurgische Intensivmedizin, Innsbruck, Tyrol
- Belgium (7):
  - Hôpital Erasme, Brussels, Brussels Capital
  - CHU UCL Mont Godinne, Yvoir, Namur
  - University Hospital Ghent, Ghent, Oost Vlaanderen
  - University Hospital Antwerpen, Antwerp
  - Cliniques Universitaires Saint Luc-UCL, Brussels
  - CHU Brugmann, Brussels
  - UZ Brussel, Brussels
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne, Brno, South Moravian
  - Oblastni nemocnice Kolin, a.s., Kolín
  - Fakultni nemocnice Plzen, Pilsen
- Finland (3):
  - Helsingin Yliopistollinen Keskussairaala, Helsinki
  - Kuopion Yliopistollinen Sairaala, Kuopio
  - Tampereen yliopistollinen sairaala, Tampere
- France (8):
  - Hôpital Universitaire Dupuytren, Limoges, Haute-Vienne
  - Hôpital Charles Nicolle, Rouen, Seine-Maritime
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon, Vendée
  - CHU Angers, Angers
  - Centre Hospitalier Victor Dupouy - hopital, Argenteuil
  - CHRU Nantes - Hospital, Nantes
  - Hôpital Lariboisière, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (7):
  - University Hospital Frankfurt, Anaesthesia, Intensive Care Medicine & Pain Therapy, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover Hospital - Zentrum Innere Medizin - Klinik fuer Pneumologie, Hanover, Lower Saxony
  - Universitätsmedizin Greifswald Klinik für Anästhesiologie, IntensivmedizinNotfallmedizin und Schmerzmedizin, Greifswald, Mecklenburg-Vorpommern
  - Universitätsklinikum Schleswig-Holstein - Klinik für Anästhesiologie und Operative Intensivmedizin, Kiel, Schleswig-Holstein
  - Helios Klinikum Erfurt -Klinik fur Anaesthesie, Intensivmedizin und Schmerztherapie, Erfurt, Thuringia
  - Universitatsklinikum Jena - Klinik für Anästhesiologie und Intensivmedzin, Jena, Thuringia
  - Universitätsklinikum Hamburg Eppendorf Department Intensive Care Medicine, Hamburg
- St. Vincent's University Hospital, Dublin, Ireland
- Netherlands (9):
  - Radboud University Nijmegen, Nijmegen, Gelderland
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - VU Medisch Centrum, Amsterdam, North Holland
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Medical Center Leeuwarden, Leeuwarden, Provincie Friesland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - Ikazia Ziekenhuis, Rotterdam, South Holland
  - Gelre Ziekenhuizen - Hospital, Apeldoorn
- Spain (7):
  - Hospital Universitario Germans Trias i Pujol Medicina Intensiva Hospital General,, Badalona, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona, Catalonia
  - Corporacio Sanitaria Parc Tauli, Sabadell, Catalonia
  - Hospital Mutua de Terrassa, Terrassa, Catalonia
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Unidad de Cuidados Intensivos Hospital General, Madrid
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
- United Kingdom (5):
  - Royal Surrey County Hospital - Intensive Care Unit, Guildford, Surrey
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal London Hospital, London
  - University College London, London
  - St James University Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pickkers P, Mehta RL, Murray PT, Joannidis M, Molitoris BA, Kellum JA, Bachler M, Hoste EAJ, Hoiting O, Krell K, Ostermann M, Rozendaal W, Valkonen M, Brealey D, Beishuizen A, Meziani F, Murugan R, de Geus H, Payen D, van den Berg E, Arend J; STOP-AKI Investigators. Effect of Human Recombinant Alkaline Phosphatase on 7-Day Creatinine Clearance in Patients With Sepsis-Associated Acute Kidney Injury: A Randomized Clinical Trial. JAMA. 2018 Nov 20;320(19):1998-2009. doi: 10.1001/jama.2018.14283. PMID 30357272
- [Derived] Peters E, Mehta RL, Murray PT, Hummel J, Joannidis M, Kellum JA, Arend J, Pickkers P. Study protocol for a multicentre randomised controlled trial: Safety, Tolerability, efficacy and quality of life Of a human recombinant alkaline Phosphatase in patients with sepsis-associated Acute Kidney Injury (STOP-AKI). BMJ Open. 2016 Sep 27;6(9):e012371. doi: 10.1136/bmjopen-2016-012371. PMID 27678541

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients suffering sepsis associated acute kidney injury and admitted to the ICU were recruited from December 2014 to May 2017 in 10 European countries and the USA.53 Sites recruited patients. Sepsis diagnosis was established following the Sepsis-2 criteria and AKI diagnosis was established following the AKIN criteria.
Pre-assignment Details: Patients should show a continuation of AKI measured by a confirmatory serum creatinine value, which did not decrease > or = 0.3 mg/dL compared to the diagnostic serum creatinine value or by a continuation of urine output of < 0.5 mg/kg/h for more than 6 hours.
Groups:
- Placebo: One hour IV infusion of Placebo once daily for three consecutive days
- 0.4 mg/kg (250 U/kg) recAP: One hour IV infusion of 0.4 mg/kg recAP once daily for three consecutive days
- 0.8 mg/kg (500 U/kg) recAP: One hour IV infusions of 0.8 mg/kg recAP once daily for three consecutive days
- 1.6 mg/kg (1000 U/kg) recAP: One hour IV infusions of 1.6 mg/kg recAP once daily for three consecutive days
Period: Overall Study
Arm/Group | Placebo | 0.4 mg/kg (250 U/kg) recAP | 0.8 mg/kg (500 U/kg) recAP | 1.6 mg/kg (1000 U/kg) recAP
Started | 116 | 39 | 35 | 111
ITTcombined (Enrolled patients randomized to study drug, excl patients randomized during IA to 2 dropped doses) | 116 | 31 | 32 | 111
ITTinterim (All randomized patients and included in the interim analysis (IA)) | 30 | 31 | 32 | 29
Safety Population (All randomized patients who received at least one dose of study drug) | 112 | 38 | 35 | 109
Completed | 71 | 25 | 24 | 81
Not Completed | 45 | 14 | 11 | 30
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 31 | 8 | 5 | 16
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 4
Not completed — different, e.g adm other hospital | 12 | 3 | 3 | 10

BASELINE CHARACTERISTICS:
Population: ITT combined population
Groups:
- Placebo: One hour IV infusion of placebo once daily for 3 consecutive days
- 0.4 mg/kg (250 U/kg) recAP: One hour IV infusions of 0.4 mg/kg recAP once daily for three consecutive days
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.4 mg/kg (250 U/kg) recAP | 0.8 mg/kg (500 U/kg) recAP | 1.6 mg/kg (1000 U/kg) recAP | Total
Number analyzed (Participants) | 116 | 31 | 32 | 111 | 290
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68.0 [61.0 to 75.0] | 67.0 [61.0 to 72.0] | 66.5 [62.5 to 72.0] | 65.0 [57.0 to 73.0] | 67.0 [59.0 to 73.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 8 | 16 | 29 | 85
  Male | 84 | 23 | 16 | 82 | 205
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 95 | 25 | 27 | 95 | 242
  Black | 4 | 0 | 0 | 1 | 5
  Asian | 1 | 2 | 0 | 1 | 4
  Other | 0 | 0 | 1 | 0 | 1
  Not collected | 16 | 4 | 4 | 14 | 38
Region of Enrollment [Number; unit: participants]
  Austria | 11 | 2 | 2 | 11 | 26
  Netherlands | 28 | 8 | 7 | 28 | 71
  Belgium | 12 | 5 | 5 | 13 | 35
  United States | 14 | 1 | 1 | 11 | 27
  Czechia | 3 | 2 | 3 | 5 | 13
  Ireland | 1 | 0 | 0 | 0 | 1
  Finland | 6 | 1 | 3 | 6 | 16
  United Kingdom | 12 | 5 | 3 | 11 | 31
  France | 16 | 4 | 4 | 14 | 38
  Spain | 9 | 3 | 4 | 7 | 23
  Germany | 4 | 0 | 0 | 5 | 9
BMI [Median (Inter-Quartile Range); unit: kg/m2] — Population: BMI is composed of weight and height measurements. For some patients no Height was available
  kg/m2
    number analyzed (Participants) | 115 | 30 | 29 | 110 | 284
    (all) | 26.3 [23.9 to 29.4] | 25.8 [22.4 to 28.4] | 27.4 [25.2 to 30.7] | 26.8 [23.9 to 30.2] | 26.6 [23.9 to 29.4]
APACHE II [Median (Inter-Quartile Range); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation II score (APACHE II) is a severity-of-disease used in adults upon admission to the ICU. A score of 0 to 71 is calculated based on 12 routine measurements and the higher scores corresponds to a more severe disease state and a higher risk of mortality. Parameters included in the score are the patient's age, AaDO2 or PaO2 (depending on FiO2), temperature (rectal), Mean arterial pressure, pH arterial, Heart rate, Respiratory rate, Sodium (serum), Potassium (serum), Creatinine, Hematocrit, White blood cell count and Glasgow Coma Scale Population: One patient did not have an APACHE score at baseline
  units on a scale
    number analyzed (Participants) | 116 | 31 | 32 | 110 | 289
    (all) | 26.0 [20.0 to 33.5] | 30.0 [25.0 to 35.0] | 26.0 [20.0 to 34.5] | 25.0 [19.0 to 31.0] | 26.0 [21.0 to 33.0]
SOFA score [Median (Inter-Quartile Range); unit: units on a scale] — Sequential Organ Failure Assessment score (SOFA score) is used to track a person's status during the stay in an intensive care unit (ICU) to determine the extent of a person's organ function or rate of failure. The SOFA score is composed of six different sub-scores, concerning respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Each of the six subscores can have a maximal score of 4. The higher the score the more severe the organ dysfunction is (SOFA score ranges theoretically from 0-30). Population: Not all patients in ITT did had a baseline SOAFA score
  units on a scale
    number analyzed (Participants) | 113 | 29 | 32 | 108 | 282
    (all) | 10.0 [8.0 to 12.0] | 10.0 [8.0 to 13.0] | 9.0 [8.0 to 11.0] | 10.0 [8.0 to 12.0] | 10.0 [8.0 to 12.0]
Mechanical ventilation [Count of Participants; unit: Participants] | 68 | 23 | 20 | 70 | 181
Vasopressor/ionotropic therapy [Count of Participants; unit: Participants] | 103 | 28 | 30 | 102 | 263
Heart rate [Median (Inter-Quartile Range); unit: beats/min] | 98.0 [85.0 to 111.0] | 93.0 [77.0 to 115.0] | 90.0 [75.5 to 107.5] | 95.0 [83.0 to 110.0] | 95.5 [81.0 to 110.0]
Bloodpressure [Median (Inter-Quartile Range); unit: mmHg] — Population: Lacking blood pressure results
  mmHg
    Systolic bloodpressure: number analyzed (Participants) | 116 | 31 | 32 | 110 | 289
    Systolic bloodpressure | 112.0 [101.5 to 131.5] | 108.0 [100.0 to 119.0] | 118.5 [96.0 to 131.0] | 107.0 [95.0 to 119.0] | 110 [98.0 to 123.0]
    Diastolic bloodpressure | 56.5 [51.0 to 63.5] | 54.0 [49.0 to 62.0] | 58.0 [54.0 to 62.0] | 55.0 [49.0 to 62.0] | 56.0 [50.0 to 62.0]
Body temperature [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 114 | 31 | 32 | 108 | 285
    <36oC | 11 | 4 | 5 | 11 | 31
    >= 36oC and =< 38oC | 76 | 20 | 22 | 79 | 197
    >38oC | 27 | 7 | 5 | 18 | 57
eGFR [Median (Inter-Quartile Range); unit: mL/min] — Population: Missing data
  mL/min
    number analyzed (Participants) | 102 | 27 | 28 | 98 | 255
    (all) | 37.5 [23.9 to 50.8] | 27.2 [20.0 to 42.4] | 25.6 [20.4 to 40.7] | 29.7 [20.5 to 46.5] | 31.8 [21.0 to 47.8]
Endogenous Creatinine clearance [Median (Inter-Quartile Range); unit: mL/min] — Population: Missing data
  mL/min
    Baseline: number analyzed (Participants) | 49 | 10 | 12 | 46 | 117
    Baseline | 31.8 [14.7 to 62.5] | 14.4 [8.8 to 58.0] | 26.0 [5.4 to 30.6] | 24.1 [10.5 to 54.9] | 27.9 [9.3 to 58.0]
    Day 1: number analyzed (Participants) | 103 | 30 | 31 | 102 | 266
    Day 1 | 35.9 [12.2 to 82.9] | 28.3 [4.3 to 64.4] | 25.2 [9.4 to 61.0] | 26.0 [8.8 to 59.5] | 29.4 [10.0 to 67.9]
AKI stage [Count of Participants; unit: Participants] — AKI stage defined 3 stages based on serum Creatinine measurements or urine output and provide a classification of the severity of the acute kidney injury (see KDIGO guidelines 2012 for more details). AKI Stage 3 being the most severe stage of kidney injury. Population: Missing data
  Participants
    AKI Stage 1: number analyzed (Participants) | 112 | 31 | 32 | 109 | 284
    AKI Stage 1 | 91 | 22 | 23 | 81 | 217
    AKI Stage 2: number analyzed (Participants) | 112 | 31 | 32 | 109 | 284
    AKI Stage 2 | 16 | 5 | 5 | 17 | 43
    AKI Stage 3: number analyzed (Participants) | 112 | 31 | 32 | 109 | 284
    AKI Stage 3 | 5 | 4 | 4 | 11 | 24
Urine output [Median (Inter-Quartile Range); unit: mL/h] — Population: Missing data
  mL/h
    number analyzed (Participants) | 53 | 13 | 14 | 50 | 130
    (all) | 60.0 [21.8 to 99.3] | 50.0 [21.7 to 101.7] | 27.4 [16.4 to 50.0] | 39.1 [10.9 to 85.7] | 46.3 [16.7 to 91.7]
Serum Creatinine [Median (Inter-Quartile Range); unit: mg/dL] — Population: Missing data
  mg/dL
    number analyzed (Participants) | 113 | 29 | 32 | 110 | 284
    (all) | 1.8 [1.3 to 2.4] | 2.3 [1.5 to 2.8] | 1.9 [1.5 to 2.8] | 2.0 [1.4 to 2.8] | 1.9 [1.4 to 2.6]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Time Corrected Endogenous Creatinine Clearance From Day 1 to Day 7 (AUC1-7)
Description: Primary endpoint is calculated as the average of the standardized endogenous creatinine clearance values over the first seven days between the placebo and 1.6 mg/kg recAP arm.
  Standardized endogenous creatinine clearance is assessed on each days from D1 to Day 7 during a 6 +/- 1 hour period and calculated in mL/min as the mean creatinine clearance over the period. The study started with 4 treatment arms of which 0.4 mg/kg recAP and the 0.8 mg/kg recAP were dropped after the interim analysis. The number of the patients in the dropped arm are respectively 30 and 32. Therefore the statistical analysis has been performed only on the placebo and 1.6 mg/kg group.
Time Frame: 7 days
Population: ITT combined includes all patients randomized in part 1 and part 2 of the study, excluding patients recruited whilst the interim analysis is performed to treatment arms not selected for Part 2. Some values were discarded by the adjudication committee.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | Placebo | 0.4 mg/kg (250 U/kg) recAP | 0.8 mg/kg (500 U/kg) recAP | 1.6 mg/kg (1000 U/kg) recAP
Number analyzed (Participants) | 106 | 30 | 32 | 108
mL/min
  Part 1: number analyzed (Participants) | 28 | 29 | 30 | 29
  Part 1 | 41.35 [19.00 to 130.15] | 43.30 [16.40 to 93.30] | 64.25 [14.20 to 104.00] | 61.10 [6.80 to 93.50]
  Part 2: number analyzed (Participants) | 77 | 0 | 0 | 80
  Part 2 | 44.51 [17.71 to 108.51] |  |  | 51.76 [17.61 to 94.58]
  Part 1 + Part 2 | 45.6 [17.7 to 112.4] | 46.95 [6.58 to 88.40] | 63.54 [8.07 to 96.77] | 55.1 [15.0 to 93.9]
Statistical Analysis 1: Comparison: Placebo vs 1.6 mg/kg (1000 U/kg) recAP; Analysis for Part 1; Test type: Superiority; p = 0.949, ANOVA; Difference in LS means = -16.53, 95% CI 2-sided [-62.57 to 29.50], Standard Error of Mean 19.243
Statistical Analysis 2: Comparison: Placebo vs 1.6 mg/kg (1000 U/kg) recAP; Analysis for Part 2; Test type: Superiority; p = 0.691, ANOVA; Difference in LS means = -4.65, 95% CI 2-sided [-23.09 to 13.80], Standard Error of Mean 9.305
Statistical Analysis 3: Comparison: Placebo vs 1.6 mg/kg (1000 U/kg) recAP; Combination of analysis results from Part 1 (see statistical Analysis 1) and Part 2 (see Statistical analysis 2); Test type: Superiority; p = 0.896, Inverse normal method; Combined p-value = 0.896 — The p-values from Part 1 (see Statistical Analysis 1) and Part 2 (see Statistical Analysis 2) were combined to an overall p-value using the inverse normal method

2. Secondary Outcome: Number of Participants Who Had Renal Replacement Therapy (RRT) During the Period Day 1 to Day 28, Inclusive
Description: During the study the days on Renal Replacement Therapy (RRT) was recorded for each patients. During the first 7 days of the study (D1 to D7 included), patients were only allowed to receive continuous RRT, thereafter patients were also allowed to receive intermittent RRT. Standardization of RRT was attempted by providing guidelines to start and stop RRT (see protocol). Statistical analysis was only performed on the placebo and 1.6 mg/kg recAP arm due to the small number of patients treated with the doses of 0.4 mg/kg and 0.8 mg/kg recAP. Those two doses were dropped in part 2 of the study.
Time Frame: 28 days
Population: ITT combined
Measure: Count of Participants; unit: Participants
Groups:
- 0.8 mg/kg (500U/kg) recAP: One hour IV infusions of 0.8 mg/kg recAP once daily for three consecutive days
Arm/Group | Placebo | 0.4 mg/kg (250 U/kg) recAP | 0.8 mg/kg (500U/kg) recAP | 1.6 mg/kg (1000 U/kg) recAP
Number analyzed (Participants) | 116 | 31 | 32 | 111
Participants | 34 | 11 | 7 | 40
Statistical Analysis 1: Comparison: Placebo vs 1.6 mg/kg (1000 U/kg) recAP; Test type: Superiority; p = 0.28, Chi-squared; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.8 to 2.4]

3. Other Pre Specified Outcome: All-cause Mortality at Day 28
Description: Number of patients in the ITT set, who died in the period between day 1 to day 28. Statistical analysis was only performed on the placebo and 1.6 mg/kg recAP arm due to the small number of patients treated with the doses of 0.4 mg/kg and 0.8 mg/kg recAP. Those two doses were dropped in part 2 of the study.
Time Frame: Day 28
Population: ITT set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.4 mg/kg (250 U/kg) recAP | 0.8 mg/kg (500 U/kg) recAP | 1.6 mg/kg (1000 U/kg) recAP
Number analyzed (Participants) | 116 | 31 | 32 | 111
Participants | 31 | 8 | 4 | 16
Statistical Analysis 1: Comparison: Placebo vs 1.6 mg/kg (1000 U/kg) recAP; Test type: Superiority; p = 0.02, Cochran-Mantel-Haenszel; Mean Difference (Net) = 0.12, 95% CI 2-sided [0.02 to 0.23]

4. Other Pre Specified Outcome: All-cause Mortality at Day 90
Description: Number of patients in the ITT set, who died in the period between Day 1 and Day 90 Statistical analysis was only performed on the placebo and 1.6 mg/kg recAP arm due to the small number of patients treated with the doses of 0.4 mg/kg and 0.8 mg/kg recAP. Those two doses were dropped in part 2 of the study.
Time Frame: Day 90
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.4 mg/kg (250 U/kg) recAP | 0.8 mg/kg (500 U/kg) recAP | 1.6 mg/kg (1000 U/kg) recAP
Number analyzed (Participants) | 116 | 31 | 32 | 111
Participants | 34 | 9 | 6 | 19
Statistical Analysis 1: Comparison: Placebo vs 1.6 mg/kg (1000 U/kg) recAP; Test type: Superiority; p = 0.03, Cochran-Mantel-Haenszel; Mean Difference (Net) = 0.12, 95% CI 2-sided [0.01 to 0.23]

5. Other Pre Specified Outcome: Number of Participants Meeting at Least One MAKE 60 Criteria
Description: Make 60 is composed of patients that meet at least one of the following criteria at day 60:
  1. had eGFR < 60 mL/min (calculated by using the CKD-EPI formula) or
  2. became dialysis dependent up to Day 60 or
  3. died prior to Day 60 Statistical analysis was only performed on the placebo and 1.6 mg/kg recAP arm due to the small number of patients treated with the doses of 0.4 mg/kg and 0.8 mg/kg recAP. Those two doses were dropped in part 2 of the study.
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.4 mg/kg (250 U/kg) recAP | 0.8 mg/kg (500 U/kg) recAP | 1.6 mg/kg (1000 U/kg) recAP
Number analyzed (Participants) | 116 | 31 | 32 | 111
Participants | 46 | 13 | 11 | 30
Statistical Analysis 1: Comparison: Placebo vs 1.6 mg/kg (1000 U/kg) recAP; Test type: Superiority; p = 0.045, Regression, Logistic; Hazard Ratio (HR) = 1.77, 95% CI 2-sided [1.0 to 3.1]

6. Other Pre Specified Outcome: Number of Patients Who Meet at Least One of the MAKE 90 Criteria
Description: Make 90 includes patients who meet at least one of the following parameters at Day 90:
  1. had eGFR <60 ml/min at Day 90, estimated by the CKD-EPI formula based on a serum creatinine or
  2. was dialysis dependent up to Day 90 or
  3. was hospitalized for a new episode of acute kidney injury prior to Day 90 or
  4. died, prior to Day 90 Statistical analysis was only performed on the placebo and 1.6 mg/kg recAP arm due to the small number of patients treated with the doses of 0.4 mg/kg and 0.8 mg/kg recAP. Those two doses were dropped in part 2 of the study.
Time Frame: Day 90
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.4 mg/kg (250 U/kg) recAP | 0.8 mg/kg (500U/kg) recAP | 1.6 mg/kg (1000 U/kg) recAP
Number analyzed (Participants) | 116 | 31 | 32 | 111
Participants | 46 | 13 | 10 | 29
Statistical Analysis 1: Comparison: Placebo vs 1.6 mg/kg (1000 U/kg) recAP; Test type: Superiority; p = 0.03, Regression, Logistic; Hazard Ratio (HR) = 1.85, 95% CI 2-sided [1.06 to 3.26]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the patient signed the informed consent form until Day 28
Arm/Group | Placebo | 0.4 mg/kg (250 U/kg) recAP | 0.8 mg/kg (500 U/kg) recAP | 1.6 mg/kg (1000 U/kg) recAP
All-Cause Mortality (participants affected / at risk) | 33/112 | 10/38 | 6/35 | 19/109
Serious Adverse Events (participants affected / at risk) | 56/112 | 18/38 | 11/35 | 47/109
Other Adverse Events (participants affected / at risk) | 111/112 | 35/38 | 31/35 | 103/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=112) | 0.4 mg/kg (250 U/kg) recAP (N=38) | 0.8 mg/kg (500 U/kg) recAP (N=35) | 1.6 mg/kg (1000 U/kg) recAP (N=109)
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium Difficile infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Iatrogenic infection (Infections and infestations) | 0 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 2
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0 | 1
Necrotising soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Peritoneal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 1 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0 | 2 | 4
Pneumonia herpes viral (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 11 | 2 | 4 | 3
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Gastrointestinal haemorrage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Intral abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ischemia enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 1 | 4
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Arterial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 4 | 0 | 1 | 4
Cardiac failure (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 0 | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardiac infarction (Cardiac disorders) | 1 | 0 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Astenia (General disorders) | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 7 | 2 | 0 | 5
Arterial haemorrhage (Vascular disorders) | 1 | 0 | 0 | 1
Arterial insufficiency (Vascular disorders) | 1 | 0 | 0 | 0
Capillary disorder (Vascular disorders) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral ischemia (Vascular disorders) | 1 | 0 | 0 | 2
Shock (Vascular disorders) | 2 | 0 | 0 | 1
Shock haemorrhage (Vascular disorders) | 1 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 1
Metabolic encepalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Neuromyopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Anastomic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic haematoma (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Caxhexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Connective tissue disorders fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=112) | 0.4 mg/kg (250 U/kg) recAP (N=38) | 0.8 mg/kg (500 U/kg) recAP (N=35) | 1.6 mg/kg (1000 U/kg) recAP (N=109)
Abdominal Pain (Gastrointestinal disorders) | 9 | 0 | 3 | 3
Constipation (Gastrointestinal disorders) | 13 | 1 | 3 | 12
Diarrhoea (Gastrointestinal disorders) | 12 | 2 | 3 | 16
Ileus apralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 7
Impaired gastric emptying (Gastrointestinal disorders) | 8 | 1 | 2 | 8
Nausea (Gastrointestinal disorders) | 14 | 4 | 3 | 13
Vomiting (Gastrointestinal disorders) | 5 | 3 | 1 | 6
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 0
Fungal infection (Infections and infestations) | 3 | 2 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 3 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 1 | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 2 | 0 | 6
Hypernatraemia (Metabolism and nutrition disorders) | 10 | 0 | 1 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 5 | 3 | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 2 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 2 | 1 | 6
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 0 | 2 | 3
Metabolic alkalosis (Metabolism and nutrition disorders) | 3 | 0 | 2 | 3
Generalised oedemia (General disorders) | 5 | 3 | 2 | 9
Multiple organ dysfunction syndrome (General disorders) | 7 | 2 | 0 | 5
Oedema peripheral (General disorders) | 17 | 4 | 5 | 21
Pain (General disorders) | 5 | 0 | 2 | 1
Pyrexia (General disorders) | 7 | 2 | 3 | 10
Arterial flutter (Cardiac disorders) | 1 | 2 | 2 | 3
Bradycardia (Cardiac disorders) | 3 | 2 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 5 | 1 | 0 | 7
Agitation (Psychiatric disorders) | 6 | 2 | 2 | 13
Anxiety (Psychiatric disorders) | 3 | 3 | 2 | 3
Delirium (Psychiatric disorders) | 20 | 5 | 5 | 14
Insomnia (Psychiatric disorders) | 10 | 2 | 2 | 13
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 4 | 14
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 10 | 2 | 6 | 14
Hypotension (Vascular disorders) | 10 | 5 | 2 | 6
Phlebitis (Vascular disorders) | 2 | 1 | 2 | 2
Blood phosphorus decreased (Investigations) | 2 | 2 | 1 | 3
Breath sound abnormal (Investigations) | 0 | 1 | 2 | 1
Cardiac murmur (Investigations) | 1 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 9 | 2 | 1 | 8
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 9
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Intensive care unit acquired weakness (Nervous system disorders) | 4 | 1 | 2 | 5
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 4 | 2 | 2 | 4
Disorientation (Psychiatric disorders) | 0 | 3 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Haematoma (Vascular disorders) | 5 | 1 | 2 | 2
Blood potassium decreased (Investigations) | 2 | 0 | 2 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT02182440/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT02182440/SAP_001.pdf